CLINICAL TRIAL: NCT02514590
Title: Multi-center, Prospective, Clinical Trial of Wireless Spinal Cord Stimulation in the Treatment of Chronic Pain
Brief Title: Wireless Spinal Cord Stimulation for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Collaborators: The Cleveland Clinic (Other); The Center for Clinical Research, Winston-Salem, NC (Other); Anesthesia Pain Care Consultants, Tamarac, FL, USA (Unknown); Precision Spine Care, Tyler, TX, USA (Unknown); Nuvo Spine and Sports Institute & Ortho Regenerative Center, Encino, CA, USA (Unknown); Compass Research LLC, Orlando, FL, USA (Unknown); USC Spine, Keck hospital of USC, Los Angeles, CA, USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30-00113
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Freedom SCS System - 1500 HZ (Experimental): Epidural Space covering vertebrae level T8-T11 determined by paresthesia mapping for painful area.
  Interventions: Device: Freedom SCS System

INTERVENTIONS:
Device: Freedom SCS System — This Freedom SCS System is based on wireless neuromodulation technology. This technology includes octapolar stimulators with embedded receivers. The energy source is a small, external, rechargeable transmitter, which is worn by the subject. The device is programmed to have a 5-1500 Hz therapy.

SUMMARY:
The purpose of this study is to assess the effectiveness of the Stimwave Spinal Cord Stimulator (SCS) System for treatment of chronic pain

DETAILED DESCRIPTION:
This is a multi-center, prospective study in which subjects will receive a Freedom SCS System and to receive stimulation at a frequency between 5 Hz to 1500 Hz . Enrollment will continue until 49 subjects have been implanted.

Subjects will have chronic back or back and leg pain refractory to standard medical treatment associated with Failed Back Surgery Syndrome (FBSS). Subjects will be followed for a 6-month period after a maximum one-month trial period. At the end of 6 months follow-up, all subjects will assess the outcomes of their appointed therapy and continue with long-term use of the system.

Stimulators will be placed at the following sites to target the painful area:

• Epidural Space midline covering vertebrae levels T8 through T11 (one stimulator placed at the top of T8 and the second stimulator placed at the middle of T9). Paresthesia mapping will be utilised to determine the optimal location for stimulation of the painful area.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at time of informed consent;
* Subjects have been diagnosed with chronic back or back and leg pain with an average VAS > 5 (on a 10 scale) over the course of the last month for back pain based on baseline pain diary;
* Subject diagnosis with chronic back or back and leg pain associated with FBSS refractory to conventional medical management for at least 12 months prior to enrollment;
* Based on the medical opinion of the Principal Investigator, subject has a stable pain medication regiment;
* Based on the medical opinion of the Principal Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;
* Based on the opinion of the Principal Investigator, subject is willing and able to operate the patient programmer, recharging equipment, diary and has the ability to undergo study assessments and provide accurate responses;
* Based on the opinion of the implanter, subject is a good surgical subject for the implant procedure;
* Subject is willing to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements;
* Subject is male or non-pregnant female;
* Subject is deemed to be neuro-psycho-socially appropriate for implantation therapies based of the assessment of a Clinical Psychologist, using face-to-face encounters and the psychological testing described in the measures;
* Subject is capable of giving informed consent;
* Subject lives within reasonable distance from the study site (circumference of 50 miles).

Exclusion Criteria:

* Obvious mechanical instability related to pain (diagnosed by imaging taken within the past 6 months);
* Unresolved Malignancies in last six months;
* Subject has post-herpetic neuralgia (shingles);
* Subject has an active systemic infection or is immune-compromised;
* Based on the medical opinion of the Principal Investigator, Psychologist and/or Psychiatrist, the subject has other psychological conditions (e.g., psychosis, suicidal ideation, borderline personality disorder, somatization, narcissism), other health conditions (e.g., substance abuse, another chronic condition requiring the regular use of opioid medication), or other legal concerns that would preclude his/her enrollment in the study or potentially confound the results of the study;
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study;
* Insulin-dependent diabetic who is not controlled through diet and/or medication (determined by the physician) or non-insulin dependent diabetic who is not well controlled through diet and/or medication;
* Bleeding complications or coagulopathy issues;
* Pregnant/lactating or not using adequate birth control;
* A life expectancy of less than one year;
* Any active implanted device whether turned off or on;
* A previous SCS experience;
* Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Pain Score | 6 Months
  A 50% reduction in VAS scores when compared to baseline.

SECONDARY OUTCOMES:
Percentage change in VAS Back from baseline | 6 Months
  The percentage reduction in VAS back pain
Percentage change in VAS Leg from baseline | 6 Months
  The percentage reduction in VAS leg pain
Oswestry Disability Index (ODI) Score | 6 Months
  The change from baseline in functionality using the ODI
Patient Satisfaction | 6 Months
  The change in satisfaction as measured by Patient Global Impression of Change
Disability Score | 6 Months
  The change in European Quality of Life 5 Dimension
Sleep Quality | 6 Months
  Frequency of sleep disturbances reported from diary
Procedure time | 7 Days post implant
  The time measured to implant the device from operative notes
Opioid Reduction | 6 Months
  The reduction in opioids as reported by patient prescription
Adverse Events | 6 Months
  The incidence of device related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Mekhail, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - Nuvo Spine and Sports Institute & Ortho Regenerative Center, Beverly Hills, California
  - USC Spine Center, Keck Hospital of USC, Los Angeles, California
  - Compass Research, Orlando, Florida
  - Anesthesia Pain Care Consultants, Tamarac, Florida
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Precision Spine Care, Tyler, Texas